CLINICAL TRIAL: NCT05108818
Title: Characterization of Humoral and Cellular Immune Responses Elicited by Influenza Vaccination in Healthy Adults
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH); Stanford University (Other); The Scripps Research Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 849398; 21-0033 (Other: DMID); 75N93021C00015 (Other Grant/Funding Number: NIAID); Institutional Funds (Other Grant/Funding Number: University of Pennsylvania)
Record Dates: First submitted 2021-10-11; First posted 2021-11-05 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Influenza, Human
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Influenza vaccination (Experimental): Adults will receive a seasonal, inactivated, quadrivalent influenza vaccine administered intramuscularly at a dose of 15 ug of HA per component, as approved by the FDA.
  Interventions: Biological: Seasonal influenza vaccine

INTERVENTIONS:
Biological: Seasonal influenza vaccine — The seasonal influenza vaccine is administered intramuscularly at a dose of 15 ug of HA per component, as approved by the FDA.

SUMMARY:
Cellular and humoral immune responses before and after seasonal influenza vaccination will be assessed. Each year, up to 100 participants will be enrolled. To study age-specific differences in immune responses, participants with various years of birth will be enrolled. The investigators hypothesize that humans with different birth years will mount antibody and cellular responses of different specificities following seasonal influenza vaccination.

DETAILED DESCRIPTION:
The investigators and others have shown that the first influenza virus someone is exposed to leaves an immunological imprint that affects antibody responses to antigenically related influenza strains later in life. Year of birth can be used to predict influenza virus exposures during the first years of life. It is possible that immune responses to influenza vaccination later in life differ between people with different birth years, depending on what virus someone was "imprinted" with. This could result in birth year differences in antibody responses upon vaccination and vaccine effectiveness. However, the effect of year of birth on the specificity of humoral and cellular immune responses elicited by influenza vaccination has not been studied in depth. In this study, the investigators will measure influenza virus cellular and humoral immune responses in individuals of different birth years before and after influenza vaccination.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of signed and dated informed consent form
2. Stated willingness to comply with all study procedures and availability for all study visits
3. Aged 18 years and older
4. In good health based on self-reported medical conditions via an online survey

Exclusion Criteria:

1. Known allergic reactions to components of the study vaccine
2. Known latex allergy
3. History of severe reactions following previous immunization with licensed or unlicensed influenza virus vaccines
4. History of GBS within 6 weeks of receipt of a previous influenza vaccine
5. Immunosuppression as a result of an underlying illness or treatment with immunosuppressive or cytotoxic drugs, or use of anticancer chemotherapy or radiation therapy within the preceding 36 months
6. Treatment with immunoglobulin or another blood product within the 3 months prior to enrollment in this study
7. Active neoplastic disease (excluding non-melanoma skin cancer or prostate cancer that is stable in the absence of therapy) or a history of any hematological malignancy ("active" is defined as having received treatment within the past 5 years)
8. Long-term (greater than 2 weeks) usage of oral or parenteral steroids, or high-dose inhaled steroids
9. Administration of an influenza vaccine within 2 months prior to enrollment
10. Known acute or chronic medical condition that, in the opinion of the investigator or appropriate sub-investigator, would render vaccination unsafe or would interfere with the evaluation of responses
11. Participation in a study that involves an experimental agent or having received an experimental agent (other than a COVID-19 vaccine) within 1 month prior to enrollment or expecting to receive another experimental agent during the study period
12. Intends to donate blood during the study period
13. Any condition that would, in the opinion of the site investigator, place the subject at an unacceptable risk of injury or render the subject unable to meet the requirements of the protocol
14. Pregnancy
15. Known human immunodeficiency virus, hepatitis B, or hepatitis C infection
16. Any condition that the principal investigator believes may interfere with successful completion of the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 700 (Estimated)
Dates: Start 2021-10-07 (Actual); Primary Completion 2027-04-01 (Estimated); Study Completion 2028-03-31 (Estimated)

PRIMARY OUTCOMES:
Effect of year of birth on neutralizing antibody titers elicited by influenza vaccination | 7 years
  Because year of birth can be used to predict the influenza viruses circulating during the first years of life, assessing antibody responses in individuals of different birth years is one way of determining how prior exposure affects immune responses to seasonal influenza vaccination and infection. The investigators will assess how antibody responses to seasonal influenza vaccination differ in individuals across multiple age groups. Baseline serum neutralizing antibodies to post-vaccination serum neutralizing antibodies against the influenza A (H1N1 and H3N2) and influenza B viral strains that are included in the quadrivalent influenza vaccine will be compared. The investigators will compare neutralizing antibody titers between groups of individuals with different birth years. Neutralizing antibody titers against the vaccine strains will be quantified by focus reduction neutralization test (FRNT) and data will be expressed as FRNT titer.

SECONDARY OUTCOMES:
Changes in serum HAI antibodies in individuals of different birth years following influenza vaccination | 7 years
  Baseline serum antibodies will be compared to those collected after vaccination to access changes in serum hemagglutination inhibition (HAI) antibodies that block virus binding to cells. Titer will be defined as the highest dilution resulting in complete inhibition of hemagglutination in the assay. The changes measured in HAI titer between pre and post vaccination will be compared among individuals of different birth years.
Differences in levels of HA stalk-binding antibodies in individuals of different birth years following influenza vaccination | 7 years
  Baseline serum antibodies will be compared to post-vaccination serum antibodies to assess differences in levels (increase or decrease) of reactive antibodies to the HA stalk of influenza viruses. Serum antibody titers will be measured by ELISA using "headless" HA to quantify serum antibodies targeting the HA stalk. Antibody titers measured in pre and post vaccination sera will be compared among individuals of different birth years. Data will be expressed as ELISA relative units.
Differences in levels of NA-binding antibodies in individuals of different birth years following influenza vaccination | 7 years
  Baseline serum antibodies will be compared to post-vaccination serum antibodies to assess changes in levels (increase or decrease) of antibodies that inhibit NA activity (NA-binding antibodies) of different influenza viruses. NA activity will be measured via an enzyme-linked lectin assay (ELLA) and the amount of serum antibody present that inhibits NA activity of different influenza strains will be quantified. These titers measured in pre and post vaccination sera will be compared among individuals of different birth years. Data will be expressed as ELLA titer.
Assessment of the frequency of circulating T follicular helper cell response to influenza vaccination in individuals of different birth years | 7 years
  Circulating T follicular helper cells (cTfh) with be assessed among peripheral blood mononuclear cells (PBMCs) collected at baseline and after vaccination. Frequencies, defined by percent increase or decrease, will be measured by flow cytometry-based assays. Measurement of the frequencies of cTfh in response to influenza vaccination will be compared among individuals of different birth years to determine the effect of year of birth on cTfh responses following influenza vaccination.
Assessment of the functionality of circulating T follicular helper cell response to influenza vaccination in individuals of different birth years | 7 years
  Circulating T follicular helper cells (cTfh) with be assessed among peripheral blood mononuclear cells (PBMCs) collected at baseline and after vaccination. Functionality, defined by expression of specific cellular markers, will be measured by flow cytometry-based assays. Measurement of the functionality of cTfh in response to influenza vaccination will be compared among individuals of different birth years to determine the effect of year of birth on cTfh responses following influenza vaccination.
Assessment of B cell responses to influenza vaccination in individuals of different birth years | 7 years
  B cells will be assessed among PBMCs collected at baseline and after vaccination. Frequencies, defined by percent increase or decrease, and clonal expansion will be measured by flow cytometry-based and high-throughput DNA sequencing assays. These metrics will be compared among individuals of different birth years to determine the effect of year of birth on B cells responses following influenza vaccination.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
Protocol and statistical analysis plan may need to be shared for publication.
Supporting Information: Study Protocol, SAP
Time Frame: At publication
Access Criteria: Per journal publication policy